CLINICAL TRIAL: NCT05484258
Title: Loneliness and Health Outcomes in the High Need Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Francis Balucan, Medical Director, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 220958
Record Dates: First submitted 2022-07-27; First posted 2022-08-02 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Anxiety; Loneliness; Depression; Alcohol Use Disorder; Utilization, Health Care
Keywords: high need population; shared medical visits; social determinants of health
MeSH Terms: conditions — Anxiety Disorders; Depression; Alcoholism; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): On baseline screen, would be screened for depression, alcohol use, and loneliness. Loneliness screen will be checked every 3 months.
- Group Medical VIsits (Active Comparator): For this arm, patients will have three visits of a shared medical visit, wherein a physician/APP will partner with a social worker to give a discussion about topics relevant to the high need population, including managing multiple medications, managing stress, and also palliative care.
  Interventions: Behavioral: Shared Medical Visit

INTERVENTIONS:
Behavioral: Shared Medical Visit — Group visit wherein physician and Social Worker, would be discussing topics relevant to the population.
  Arms: Group Medical VIsits

SUMMARY:
The high need population are patients who have three or more chronic diseases and have a functional limitation in their ability to take care for themselves. Investigators aim to understand the effects of a support group intervention, with the use of group medical visits and understand longitudinal effects in emotional wellbeing and loneliness.

DETAILED DESCRIPTION:
The high need population with functional limitations are patients who have three or more chronic diseases and have a functional limitation in their ability to care for themselves (such as bathing or dressing) or perform routine daily tasks. Two-thirds of the population is female, and three-quarters of them are white non-Hispanic and half of the population were described as low income. The High Need Population with functional limitations also utilizes the emergency department at twice the rate of adults with multiple chronic diseases and more than three times more likely to be hospitalized than adults of other populations.

Loneliness is seen as a significant independent risk factor for poor health behaviors, physical health problems and psychiatric conditions. Loneliness and isolation are becoming a more recognized entity that contributes to worsening depression.

Investigators aim to compare the of effects of a Social Worker and Physician/APP-led support group intervention on loneliness at 9 months, after up to 3 group visits.

Shared Medical Visits as a form of support Group increase clinician-patient contact time and provide patients with support and prevention of chronic conditions increasing patient empowerment.

ELIGIBILITY:
Inclusion Criteria:

Patients who are enrolled into the VIC program. These are patients that are 18 years old and above, and have either

* HCC Score 3.0 and above
* HCC 2.0 - 3.0 and 2 or more unplanned admissions in last 12 months
* HCC 0.24 - 0.35 + ESRD OR
* Charlson Score >3, or LACE >30

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Loneliness from Baseline at 0 and at 3, 6 and 9 months. | 0, 3, 6, and 9 months
  Using the Validated De Jong Giervald Loneliness Scale, scored from 0 (not lonely) to 11 (severely lonely),

SECONDARY OUTCOMES:
Change in the number of ED visits, Inpatient, Observations | 0, 3, 6 and 9 months
  ED Visits and Hospital Utilization (Inpatient, Observation Admissions)
Change in Depression from Baseline (0), and at 3, 6, and 9 months | 0, 3,6, and 9 months
  Will be using PHQ 9 to evaluate depression in the population, 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression
Change in Active alcohol use disorders (including alcohol abuse or dependence) from Baseline (0), and at 3, 6, and 9 months | 0,3,6, and 9 months
  he AUDIT-C has 3 questions and is scored on a scale of 0-12. Each AUDIT-C question has 5 answer choices valued from 0 points to 4 points. In men, a score of 4 or more is considered positive, optimal for identifying hazardous drinking or active alcohol use disorders. In women, a score of 3 or more is considered positive. Generally the higher the score, the more likely it is that a person's drinking is affecting his or her safety.

CONTACTS AND LOCATIONS:
Overall Officials: FRANCIS S BALUCAN, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: July 2023 available for 1 year

DOCUMENTS (2):
  • Study Protocol (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT05484258/Prot_000.pdf
  • Informed Consent Form (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT05484258/ICF_001.pdf